CLINICAL TRIAL: NCT05381220
Title: The Effects of Early Mobilization in Stroke Patients on Functional Status, Psychological Distress, and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202202035RINC
Record Dates: First submitted 2022-04-24; First posted 2022-05-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2023-04

CONDITIONS: Stroke, Acute
Keywords: stroke; early mobilization
MeSH Terms: conditions — Stroke | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early mobilization in stroke patients (Experimental): Participants in the intervention group commenced early mobilization (EM) within 24-48 hours after stroke onset. The structured program included progressive bed mobility, sitting, standing, and ambulation activities, with intensity and duration adjusted according to each patient's tolerance and neurological stability. Each session lasted approximately 30 minutes, performed once or twice daily, five days per week, and continued until hospital discharge. All sessions were conducted under the supervision of trained rehabilitation nurses and physiotherapists, with progression allowed only when vital signs were stable and no neurological deterioration was observed.
  Interventions: Other: early mobilization
- usual care in stroke patients (No Intervention): Participants will receive routine rehabilitation once daily, consisting of 20 minutes of bed exercises, including both active and passive joint movements.

INTERVENTIONS:
Other: early mobilization — Patients will receive early mobilization measures within 24 to 48 hours after the onset of stroke.
  Arms: early mobilization in stroke patients

SUMMARY:
This study aims to investigate the effects of an early mobilization intervention in improving functional status, psychological distress, and quality of life in stroke patients. We hypothesize that this intervention method can significantly alleviate patient anxiety and depression, thereby promoting functional recovery and enhancing overall quality of life. Through this research, we hope to provide stroke patients with more effective exercise programs to help them regain health and well-being.

DETAILED DESCRIPTION:
This study employs an experimental design conducted on patients in the stroke unit of the hospital who are over 20 years old and have either ischemic or hemorrhagic stroke with stable vital signs post-stroke onset, limb muscle strength greater than 3 points, and good communication skills in Chinese and Taiwanese, or they can read Chinese. Eligible participants are divided into an experimental group and a control group. All participants receive standard stroke unit care, while the intervention group additionally undergoes a 3-day activity protocol. The primary and secondary outcomes are assessed at baseline and at 1, 4, and 12 weeks post-stroke. Finally, the study analyzes the effect of early intervention on improving the prognosis of stroke patients.

The data collected in this study, whether in paper form or electronically, will be documented on a computer. After completing the research report, any recordings and paper documents will be destroyed. Once the data is documented, identifiable patient information will be removed, and each record will be assigned a unique code, making individual data unidentifiable.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 20 years old.
* Patients diagnosed with infarct or hemorrhagic stroke 24 to 48 hours later. -Patients with stable vital signs, systolic blood pressure between 140- 220mmHg, heartbeat 40-130bpm, blood oxygen >92%.
* The muscle strength of the limbs is greater than 3 points.
* Can communicate in Chinese and Taiwanese.

Exclusion Criteria:

* Patients with severe mental illness, critically ill patients and cognitive dysfunction.
* Surgery patients, aphasia patients.
* NIHSS greater than 16 points for severe stroke

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Assess changes in functional status | Data were collected at three measurement time points: baseline, the fourth week, and the 12th week after stroke.
  Functional status was assessed by Barthel Activity Daily Index (BI) and modified Rankin scale (mRS) were applied to assess activities of daily life with stroke patients. The BI is consisting of 10 common activities of daily living activities. Eight of the ten items represent activities related to personal care; the remaining 2 are related to mobility. A total score out of 100; the higher the score, the greater the degree of functional independence. The mRS scale runs from 0-6, the score of 0 is no disability, 5 is disability requiring constant care for all needs, and 6 is death.
Assess changes in sychological distress | Data were collected at three measurement time points: baseline, the fourth week, and the 12th week after stroke.
  Psychological distress was measured using the Hospital Anxiety and Depression Scale (HADS) scale. It consists of 14 items, which can be divided into two subscales of seven items each: the anxiety subscale (HADS-A) and the depression subscale (HADS-D). The total HADS score was ranged from 0 to 21. A score greater than or equal to 11 indicates that the patient has anxiety or depression.

SECONDARY OUTCOMES:
Assess changes in quality of life | Data were collected at three measurement time points: baseline, the fourth week, and the 12th week after stroke.
  Quality of life was assessed using the Stroke Impact Scale (SIS) Version 3.0, which contains 59 items covering eight domains, including strength, memory and thinking, emotion, communication, activities of daily living/instrumental activities of daily living (ADL/IADL), mobility, hand function, and participation, plus one recovery item. Each domain is scored from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao Lan Wang, University, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Taipei County

IPD SHARING:
Plan to Share IPD: No